CLINICAL TRIAL: NCT01351883
Title: Peri-operative Usage of Enteric Immune-nutrition Formula (ANOM®) Versus Standard Formula for Patients Received Major Upper Gastrointestinal Surgery
Brief Title: Enteric Immune-nutrition Formula (ANOM®) for Patients Receiving Major Upper Gastrointestinal Surgery
Acronym: ANOM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Benjamin Hsieh/ Product manager, Taiwan Otsuka Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HR-98-089
Record Dates: First submitted 2011-01-31; First posted 2011-05-11 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Chronic Upper Gastrointestinal Hemorrhage
Keywords: immunomodulating diet; postoperative infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Standard enteral nutrition supplement (No Intervention): regular standard enteral nutrition(SEN) was made by hospital for patient
  Interventions: Dietary Supplement: ANOM

INTERVENTIONS:
Dietary Supplement: ANOM — the ANOM was given 800ml per day before operation, and added from POD2 to POD 14 gradually from 400ml to 1200ml

SUMMARY:
Perioperative usage of immunonutrition (ANOM®) can attenuate the pro-inflammatory cytokines and reduce postoperative infectious complications and length of hospital stay after major upper gastrointestinal surgery.

(ANOM®)immunonutrition product name

DETAILED DESCRIPTION:
Background: Perioperative usage of immunonutrition can attenuate the pro-inflammatory cytokines and reduce postoperative infectious complications and length of hospital stay after major upper gastrointestinal surgery. The aim of this study was to elucidate the effect of immunomodulating diets, ANOM®, on surgical outcome in elective major upper gastrointestinal tract operations.

Material and Methods:

Design: Prospective, randomized, controlled trial. Participants: Seventy upper gastrointestinal tract cancer patients planned to undergo major upper gastrointestinal surgery in eesophagus、stomach、pancreas or duodenum, Interventions: Patients will be divided randomly into two groups to receive ANOM® or standard diet. Before surgery, 800ml ANOM® or standard diet (SEN) will be given for 5 days by mouth. After operation, 5% Distill water (D5W) combined with ANOM® or standard diet since the 2nd post-operation day (POD2) until day 14 (POD14) or until discharged day by enteric route using nasogastric tube(NG) tube or jejunostomy. Postoperative parenteral nutrition will be given to maintain adequate nutrition.

Clinical Assessment: The preoperative and postoperative immunological parameters, infection complications, and hospital stay will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged from 18 to 80 years old
2. Patients with upper gastrointestinal diseases, and was planning to receive elective major upper gastrointestinal tract surgery, such as subtotal gastrectomy, proximal gastrectomy, total gastrectomy, esophagectomy, pancreatectomy, pancreaticoduodenectomy, duodenectomy, etc.
3. Patient is able to understand the requirements of the study and signs the Informed Consent Form.

Exclusion Criteria:

1. Patient with severe malnutrition condition, albumin < 2.6mg/ml
2. Patient with severe pulmonary, cardiovascular, renal or hepatic disease
3. Patient with immunosuppressive therapy or immunological disease recently
4. Patient with on-going infection with any condition
5. Patient with emergency operation
6. Patient with widespread metastatic disease before surgery
7. Patient with bowel obstruction disease
8. Investigator judges as subjects to be inappropriate for the clinical study (e.g., patient with severe complications)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
postoperative infectious complication | POD 14 or discharged day
  we want to evaluate the effect of ANOM on postoperative infectious complication after early feeding with ANOM

SECONDARY OUTCOMES:
immunological parameters | POD 14 or discharged day
  we want to compare the immunological parameters, IL-6, with stand diet group
Free radicles -TBARS | POD 14 or discharged day
  we will esitimate the difference blood level of free radicles by ELISA and compared with that in the standard diet group
immunological parameters | POD14 or discharged day
  we will compare the immunological parameters, IL-8, with the stand diet group.
immunological parameter | POD14 or discharged day
  We will compare the immunological parameter, IL-1, with the standard diet group
immunological parameter | POD14 or discharged day
  We will compare the immunological parameter, IL-10, with the standard diet group
immunological parameters | POD14 or discharged day
  We will compare the immunological parameter, TNF-a, with the standard diet group

CONTACTS AND LOCATIONS:
Overall Officials: Yan-Shen Shan, MD, PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (2):
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan, Taiwan
  - Department of Surgery, Tainan Hospital, Department of Health, Executive Yuan, Tainan, Taiwan